CLINICAL TRIAL: NCT05588791
Title: Pertinence de la PREscription du Scanner Corps-Entier Aux Urgences : un Outil d'Identification Des Patients à Bas Risque
Brief Title: Relevance of Whole-body Computed Tomography Prescription in the Emergency Department : an Identification Tool for Low Risk Patients
Acronym: PRE-SCEAU
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/0425/HP
Record Dates: First submitted 2022-10-14; First posted 2022-10-20 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: whole-body computed tomography — whole-body computed tomography prescription in the emergency department : an identification tool for low risk patients

SUMMARY:
The whole-body scanner (SCE) is a powerful examination that guides the management of patients severely traumatized. However, the systematic use of this examination in emergency departments is responsible for a large proportion of normal examinations. In addition to the non-negligible direct cost, the average irradiation of 20 mSv would give an adult a 1 in 1000 risk of developing a cancer. The Vittel score makes it possible to categorize pre-hospital patients as seriously traumatized to guide the sending of resources and direct them to a center equipped with a suitable technical platform.

The use of this score to condition the prescription of the ECS is at the origin of an over-triage important since one out of two patients who validates at least one criterion has no lesion on imaging. The purpose of this research project is to validate a decision support tool to objectively guide the emergency physician in its use of the ECS. At the same time, the economic impact of such a procedure will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient undergoing an SCE as part of a post-traumatic lesion assessment during a stay in the emergency room.
* Mechanism of injury: road accident or fall.
* Patient having read and understood the information letter and given his oral consent.

Exclusion Criteria:

* Neurological impairment defined by a Glasgow score of less than 8.
* Respiratory failure with SpO2 < 90% on oxygen or with the use of ventilatory assistance.
* Hemodynamic failure with vascular filling greater than 1000 cc or recourse to catecholamines.
* Acute alcoholism.
* Taking narcotics.
* History of cognitive disorders.
* Current pregnancy.
* Suicidal patient.
* Trauma related to a brawl
* Penetrating trauma.
* Hemophilia.
* Known thrombocytopenia at the time of inclusion.
* Heart, lung, liver or kidney transplant patient.
* Person deprived of liberty by an administrative or judicial decision or person placed under legal safeguard / sub-tutorship or curatorship.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients consulting in the emergency room after a trauma whose mechanism of injury is a fall or a road accident and indicated for the realization of a whole body scanner.
Sampling Method: Probability Sample
Enrollment: 2018 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
PHASE I: Assess the negative predictive value of a 15-criteria score to exclude the traumatized patient from a whole-body CT (SCE) imaging strategy to emergencies. | through study Phase 1 completion, an average of 1 year
  The main judgment criterion is defined by the uselessness of the whole body scanner, evaluated from the SCE voucher which will contain the 15 criteria from phase I.
PHASE II: To quantify the effective reduction in SCE requests after the validated score is made available on the SCE prescription vouchers. | through study Phase 2 completion, an average of 1 year
  The main judgment criterion is the prescription of an irrelevant whole-body scanner (a patient whose 15 safety criteria are validated).

CONTACTS AND LOCATIONS:
Locations (1):
- Services des Urgences Adultes, Rouen, France

IPD SHARING:
Plan to Share IPD: No